CLINICAL TRIAL: NCT00468468
Title: Mentor Integration Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2003-192; 1P50CA09817-01A1
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: CHESS and Cancer Mentor; CHESS Only; Mentor Only; Control (Internet Only)
Keywords: breast cancer; Internet; computer; support; information; education
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- CHESS Condition (Experimental): Subjects who receive the CHESS (Comprehensive Health Enhancement Support System)
  Interventions: Behavioral: CHESS (Comprehensive Health Enhancement Support System) and Human Cancer Mentor
- Mentor Condition (Experimental): Subjects who receive access to a Human Cancer Mentor only
  Interventions: Behavioral: CHESS (Comprehensive Health Enhancement Support System) and Human Cancer Mentor
- CHESS + Mentor (Experimental): Subjects who receive the CHESS system plus a Human Cancer Mentor
  Interventions: Behavioral: CHESS (Comprehensive Health Enhancement Support System) and Human Cancer Mentor
- Internet Only (No Intervention): Subjects receive routine care and nothing else

INTERVENTIONS:
Behavioral: CHESS (Comprehensive Health Enhancement Support System) and Human Cancer Mentor — computer based education and support
  Arms: CHESS + Mentor; CHESS Condition; Mentor Condition

SUMMARY:
Mentor Integration Project

This study will investigate the benefits of CHESS, a Human Cancer Mentor and the potential additional benefit of combining CHESS and a Cancer Mentor compared to Internet access for women diagnosed with breast cancer. Our goal is to advance interactive cancer communication systems, thus improving quality of life for patients and families facing cancer, especially underserved populations.

Primary Aims:

* Determine if the Internet, CHESS, a Cancer Mentor, or a combination of CHESS and the Cancer Mentor improve quality of life for women with breast cancer
* Determine which of the above conditions is most effective
* Determine which of the above conditions is most cost efficient

ELIGIBILITY:
Inclusion Criteria:

Eligibility for this protocol is as follows:

* All subjects must be within 2 months of their primary breast cancer diagnosis,
* All subjects must be at least 18 years of age,
* All subjects must be able to read and write English at the 6th-grade level
* Not homeless

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2003-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Patient quality of life | throughout study

SECONDARY OUTCOMES:
Self efficacy | throughout study
Emotional well being | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hawkins, PhD., Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Hartford Hospital, Hartford, Connecticut
  - M.D. Anderson, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin